CLINICAL TRIAL: NCT03497741
Title: Predictive Value of Procalcitonin for Bacteremia in the ICU
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0877
Record Dates: First submitted 2018-03-28; First posted 2018-04-13 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sepsis; Procalcitonin
Keywords: Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: procalcitonin measurement — For each patient were blood cultures were taken, a procalcitonin level was determined

SUMMARY:
Association between plasma procalcitonin levels and positive blood cultures in critical illness patients in the ICU.

DETAILED DESCRIPTION:
Rationale: Association of procalcitonin levels and blood cultures in critical illness patients on the ICU.

Objective: Procalcitonin is an acute phase protein. As part of the acute phase response, procalcitonin is produced during sepsis. Previous research shows that procalcitonin is a biomarker for bloodstream infection. However, there is still little known about the value of procalcitonin in diagnostics for micro-organism underlying a sepsis in ICU patients. In modern practice, blood cultures are taken when a patient is septic to determine the responsible micro-organism. When procalcitonin is a predictive value for bacteremia in the ICU, the number of blood cultures can be reduced.

Study design: An observational cohort study intervention: for each patient in the ICU blood cultures were taken, the procalcitonin level was determined. During 6 months 150 patients will be included.

Main study parameters/endpoints: this study will examine the predictive value of procalcitonin in blood cultures on the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Age > 18 years

Exclusion Criteria:

* Hemodialysis/ Continuous Veno-Venous Hemofiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU whom blood cultures are taken for suspected bacterial infection.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The predictive value of procalcitonin in blood cultures on the ICU | 6 months
  This study will examine the predictive value of procalcitonin on blood cultures on the ICU. A high value of procalcitonin is a predictor for bacteremia.
  The predictive value: procalcitonin. Primary outcome: bacteremia .

CONTACTS AND LOCATIONS:
Overall Officials: H.J. van Leeuwen, Study Chair — Rijnstate Hospital
Locations (1):
- Rijnstate hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided